CLINICAL TRIAL: NCT01457053
Title: A Randomized Controlled Pilot Study for Assessment of Coronary Flow Reserve With Cardiac PET Imaging in Acute Decompensated Heart Failure Patients Treated With Diuretics Versus Ultrafiltration
Brief Title: Assessment of Coronary Flow Reserve in Heart Failure Patients After Ultrafiltration Versus Diuretics
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Population not available for enrollment
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Myron C. Gerson, MD, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 11051904
Record Dates: First submitted 2011-10-19; First posted 2011-10-21 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Acute decompensated heart failure; Myocardial blood flow; Coronary flow reserve; Ultrafiltration; Diuretics
MeSH Terms: interventions — Sodium Potassium Chloride Symporter Inhibitors; Furosemide; Torsemide; Bumetanide; Ultrafiltration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrafiltration (Active Comparator): Patients with acute decompensated heart failure will be randomized to either ultrafiltration or diuretics (loop diuretics: furosemide, bumetanide, and/or torsemide). Patients in this arm are randomized to ultrafiltration.
  Interventions: Other: Ultrafiltration
- Diuretic Therapy (Active Comparator): Patients with acute decompensated heart failure will be randomized to either ultrafiltration or diuretic therapy ((loop diuretics: furosemide, bumetanide, and/or torsemide). The myocardial blood flow of patients treated with ultrafiltration will be actively compared to diuretic therapy with either furosemide, bumetanide, and/or torsemide.
  Interventions: Drug: Loop diuretics (furosemide, torsemide, bumetanide)

INTERVENTIONS:
Drug: Loop diuretics (furosemide, torsemide, bumetanide) — Patients with ADHF and hypervolemia will be enrolled in a prospective, randomized fashion.
  Subjects will be randomized with a computer generated random number function to either ultrafiltration or diuretic therapy within 24 hours of hospitalization for the management of fluid overload.
  Patients randomized to diuretic therapy will be treated with intravenous loop diuretics (e.g. furosemide, bumetanide, torsemide). The selection of diuretic, dose and frequency of diuretic administration will be determined by the treating physicians based upon clinical assessment of volume status, response to medication, and perceived safety.
  Other Names: Lasix, furosemide; Bumex, bumetanide; Demadex, torsemide
  Arms: Diuretic Therapy
Other: Ultrafiltration — Subjects will be randomized with a computer generated random number function to either ultrafiltration or diuretic therapy within 24 hours of hospitalization or outpatient heart failure clinic for the management of fluid overload. If randomized to the ultrafiltration arm, on admission to the hospital patients will be initiated on ultrafiltration therapy for 2-5 days.
  Patients randomized to UF will be treated using the Aquadex System 100 ultrafiltration device (CHF Solutions, Minneapolis, MN). The selection of ultrafiltration rate (fluid removal rate)will be determined by the treating physicians based upon clinical assessment of volume status and perceived safety.
  Other Names: Aquadex System 100 ultrafiltration device
  Arms: Ultrafiltration

SUMMARY:
The purpose of this research study is to compare the effects (good and bad) of ultrafiltration treatment with standard intravenous (in your vein) diuretic therapy (furosemide, torsemide, bumetanide) on your heart function and blood flow.

DETAILED DESCRIPTION:
The standard of care to treat congestive heart failure is with a class of medication called diuretics, which remove the extra fluid from the body through urination. Another way to remove extra fluid in patients with heart failure is called ultrafiltration. Ultrafiltration may result in more rapid removal of excess fluid and more rapid improvement in your symptoms compared to standard diuretic treatment. Currently, it is unknown what effects these therapies (diuretics or ultrafiltration) have on the small blood vessels in your heart. These small blood vessels are important to supply blood and oxygen to your failing heart. Thus, the purpose of this research study is to compare the effects (good and bad) of ultrafiltration treatment with standard intravenous (in your vein) diuretic therapy on your heart function and blood flow.

ELIGIBILITY:
Inclusion Criteria:

* males and non-pregnant female patients over 18 years admitted to the hospital or treated in an outpatient heart failure clinic with the primary diagnosis of acute decompensated heart failure.
* evidence of fluid overload more than 8 kg above their dry weight, and conforming to definition of hypervolemia (at least two of the following findings: more than 1+ pitting edema of the lower extremities, jugular venous pressure more than 10 cm water, pulmonary edema or pleural effusion on chest radiograph consistent with ADHF, ascites, paroxysmal nocturnal dyspnea, or equal or more than 2 pillow orthopnea.

Exclusion Criteria:

* acute coronary syndrome
* documented ischemic cardiomyopathy
* atrial fibrillation
* serum creatinine more than 3.0 mg/dL
* systolic blood pressure less than 90 mmHg
* hematocrit > 45%
* clinical instability likely to require intravenous vasopressors and/or intravenous vasoactive drugs (such as milrinone, dobutamine, nitroglycerin or nesiritide) during the present hospitalization
* severe pulmonary hypertension or use of pulmonary hypertension drugs (such as sildenafil, bosentan or other endothelin inhibitors)
* patients with documented hypertrophic obstructive cardiomyopathy or restrictive cardiomyopathy,
* patients with severe valvular heart disease,
* patients with recent cocaine use (within one month of presentation)
* patients with heart transplant
* patients with systemic infection
* patients on hemodialysis
* inability to obtain venous access
* contraindications for anticoagulation
* unable to lie flat for at least 20 minutes
* pregnant and breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron Gerson, MD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - University of Cincinnati/University Hospital, Cincinnati, Ohio
  - University Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with acute decompensated heart failure
Groups:
- Ultrafiltration: Patients with acute decompensated heart failure will be randomized to either ultrafiltration or diuretics. The myocardial blood flow of patients treated with ultrafiltration will be actively compared to diuretic therapy.
  Ultrafiltration: Subjects will be randomized with a computer generated random number function to either ultrafiltration or diuretic therapy within 24 hours of hospitalization or outpatient heart failure clinic for the management of fluid overload. If randomized to the ultrafiltration arm, on admission to the hospital patients will be initiated on ultrafiltration therapy for 2-5 days.
  Patients randomized to UF will be treated using the Aquadex System 100 ultrafiltration device (CHF Solutions, Minneapolis, MN). The selection of ultrafiltration rate (fluid removal rate)will be determined by the treating physicians based upon clinical assessment of volume status and perceived safety.
- Diuretic Therapy: Patients with acute decompensated heart failure will be randomized to either ultrafiltration or diuretic therapy. The myocardial blood flow of patients treated with ultrafiltration will be actively compared to diuretic therapy.
  Loop diuretics (furosemide, torsemide, bumetanide): Patients with ADHF and hypervolemia will be enrolled in a prospective, randomized fashion.
  Subjects will be randomized with a computer generated random number function to either ultrafiltration or diuretic therapy within 24 hours of hospitalization for the management of fluid overload.
  Patients randomized to diuretic therapy will be treated with intravenous loop diuretics (e.g. furosemide, bumetanide, torsemide). The selection of diuretic, dose and frequency of diuretic administration will be determined by the treating physicians based upon clinical assessment of volume status, response to medication, and perceived safety.
Period: Overall Study
Arm/Group | Ultrafiltration | Diuretic Therapy
Started | 2 | 2
Completed | 1 | 1
Not Completed | 1 | 1
Not completed — Unable to undergo selected treatment | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: 2 subjects completed the study. 2 subjects did not complete either arm and did not have usable data.
Arm/Group | All Study Participants
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Blood Flow
Description: Evaluate the effects of ultrafiltration (UF) compared to intravenous diuretic therapy on myocardial blood flow (MBF) and coronary flow reserve (CFR), as assessed by positron emission tomography (PET), in patients with acutely decompensated heart failure (ADHF).
Time Frame: 1 - 5 days
Population: No data analyzed due to inadequate enrollment.
Arm/Group | Ultrafiltration | Diuretic Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ultrafiltration | Diuretic Therapy
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes